CLINICAL TRIAL: NCT02436720
Title: Performance of Upper Limb (PUL) in Duchenne Muscular Dystrophy
Brief Title: Upper Limb Assessment in Duchenne Muscular Dystrophy
Acronym: PUL in DMD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Bambino Gesù Hospital (Unknown); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Azienda Ospedaliera San Giovanni Battista (Other); University of Messina (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); University of Naples (Other); IRCCS Fondazione Stella Maris (Other); Istituto Giannina Gaslini (Other); University of Padova (Other); Maggiore Bellaria Hospital, Bologna (Other); IRCCS Eugenio Medea (Other); Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other)
Responsible Party: Principal Investigator, Eugenio Mercuri, Professor of Pediatric neurology, Catholic University of the Sacred Heart
Other Study IDs: UCSCPUL
Record Dates: First submitted 2015-04-30; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The literature on outcome measures assessing upper limbs in Duchenne muscular dystrophy (DMD) is quite scanty. While there have been considerable advances for ambulant DMD boys, no prospective study has so far been devoted to outcome measures in non ambulant patients, with increasing complaints from families and patients. This information appears to be highly important not only for a better understanding of the progression of the disease but also for possible enrollment of patients in future trials.

The aim of this project is to identify outcome measures for non ambulant patients in an Italian population of DMD patients. At least 200 non ambulant DMD boys and adults will be included in the study. All patients will be assessed using the newly developed Performance of Upper limb (PUL) test. This measure will be used at baseline and 6 and 12 months after baseline. This will allow to monitor possible changes over time and the rate of changes in patients with different level of ability and age. As part of this study the investigators will also correlate possible changes in upper limb function with other measures of care and function such as the EK scale.

The investigators aim to assess the suitability of the individual measures in a large number of patients, trying to establish whether whole scales or individual items appear to be relevant across ages and level of abilities. The investigators also aim to assess the suitability of the selected measures in a multicentric setting and the quantity of training required The data collected will also be analysed using Rasch analysis in order to improve the statistical properties of the measures used.

DETAILED DESCRIPTION:
This is a multicentric study involving a large number of patients that could not be collected in a single Unit.

The aim of the project is to collect a large number of patients that will allow to assess the suitability of different measures assessing upper limb function. As DMD is a relatively rare condition, such goal can only be reached in a multicentric setting. All the participating centres (Rome Gemelli, Messina, Rome Bambin Gesù, Pavia, Genoa, Naples, Turin, Bologna, Padua, Milan, Bosisio Parini, Pisa) have a good record of cooperation in similar projects having already been involved in the validation of the North Star in DMD and of the Hammersmith Functional motor Scale for SMA.

The projects will be developed through different steps, related to different specific aims:

1. Interobserver reliability/quality and quantity of training One of the aims of the study is to assess reliability of the selected measures in a multicentric setting and the quantity of training required to be sure of the reliability among observers after the training sessions. Following our experience in the training of the North Star Ambulatory Assessment (NSAA) in the same network, the investigators have become aware that a single training session may not be sufficient to be sure that interobserver reliability will be maintained after the training sessions (Mazzone et al, 2009).
2. Natural history data collection The PUL will be applied to the whole cohort with repeated assessments at 6, 12, 18 and 24 months . This will allow to monitor possible changes over time and the rate of changes in patients with different level of ability and age. This will also help to evaluate the responsiveness to change and the level of sensitivity of the measure over an interval that would be useful for a study of a putative agent that could improve muscle power.
3. Correlation with other measures Another aim of the study is to relate possible changes in upper limb function with other measures of care and function such as the EK scale, that provides information on aspects of function, such as transfer or self feeding that are important in everyday life. Correlation with respiratory function will also be performed.
4. improving statistical properties of the scales. There has been increasing evidence in the last few years that Rasch analysis may help to improvethe statistical properties. The data collected will offer the opportunity to perform these new psychometric techniques.

ELIGIBILITY:
Inclusion Criteria:

* proven DMD

Exclusion Criteria:

* severe mental retardation

Ages: 4 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys and adults affected by Duchenne muscular dystrophy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
assessment of upper limb (PUL) | 2 years
  the test evaluates performance of upper limbs by providing a score for shoulder, elbow and distal domain and total score

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Mercuri, MD, PhD, Principal Investigator — Catholic University
Locations (1):
- Catholic University, Rome, Italy